CLINICAL TRIAL: NCT00493467
Title: Phase II Study of Zevalin for the Treatment of Early-Stage Indolent Lymphomas
Brief Title: Zevalin (Ibritumomab Tiuxetan) for Early Stage Indolent Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Biogen (Industry); CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0512; NCI-2012-01569 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Lymphoma; Indolent Lymphomas; Ibritumomab Tiuxetan; Zevalin
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zevalin (Experimental): Ibritumomab Tiuxetan (Zevalin) + Rituximab
  Interventions: Drug: Ibritumomab Tiuxetan (Zevalin); Drug: Rituximab

INTERVENTIONS:
Drug: Ibritumomab Tiuxetan (Zevalin) — 111In Zevalin (5 mCi of ^111In, 1.6 mg of Ibritumomab Tiuxetan) Intravenously Over 10 minutes on Day 1.
  90Y Zevalin 0.3 or 0.4 mCi/kg Intravenously Over 10 minutes on Day 8.
  Other Names: Ibritumomab; Zevalin; IDEC-Y2B8
Drug: Rituximab — 250 mg/m^2 Intravenously Over 4-6 Hours On Days 1 and 8.
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to find out if giving (Rituxan) rituximab with 90Y (ibritumomab tiuxetan) (90 Y Zevalin®) may be effective in treating low-grade lymphoma. The safety of this combination treatment will also be studied.

DETAILED DESCRIPTION:
90 Y Zevalin and rituximab are both designed to attach to lymphoma cells, causing them to die.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a physical exam. Blood (about 2 to 3 teaspoons) and urine will be collected for routine tests. You will have a chest x-ray and computerized tomography (CT) scans of the neck, chest, abdomen (stomach area), and pelvis.

A PET scan is also recommended. A PET (Positron Emission Tomography) scan is a medical technique that monitors the activity in the brain and other organs by tracking the movement of a special radioactive solution through the body. The radioactive solution is either inhaled as a mist or injected into a vein. The radioactive solution is usually made from simple sugar that has radioactive particles attached to it. After the solution is injected into a vein or inhaled, the PET scanner takes pictures of the radioactive solution as it moves through the body and collects in various organs. By watching how the solution travels through the body and studying where the solution collects, researchers can learn the extent of disease in certain organs in the body.

You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). You will have a bone marrow aspirate and biopsy performed. To collect a bone marrow aspirate and biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found to be eligible to take part in this study, you will be given diphenhydramine (Benadryl) by vein and you will take acetaminophen (Tylenol) by mouth before each dose of rituximab. This is done to help decrease the risk of developing side effects of rituximab. You will then receive 1 dose of rituximab by vein over about 4-6 hours on Day 1 of treatment. After treatment with rituximab, you will then be given 111 In Zevalin (this is a radioactive agent that binds to rituximab to help with imaging exams), by vein over about 10 minutes. This is so researchers can use a special camera to see where the drug is in your body.

You will have imaging performed (on a camera, like an x-ray) on either Day 2 or 3. On Day 8 (7 days after the first dose of rituximab) you will receive a second dose of rituximab. You will also be given Benadryl, Tylenol, and 90Y Zevalin in the same manner as on Day 1.

If you experience intolerable side effects while on this study, you may be removed from this study. Your treatment on the study will end on Day 8.

You will return for follow-up tests for 4 years. Blood (about 2 tablespoons) will be drawn weekly for the first 3 months. Blood (about 2 tablespoons each time) will also be drawn at month 6 and 9 of the first year, and every 6 months in the second, third, and fourth years. You may also have CT scans, PET scans (which are recommended), x-rays, and bone marrow biopsies and aspirates performed, if your doctor thinks they are necessary.

Your participation on this study will end in about 4 years.

This is an investigational study. 90 Y Zevalin and rituximab are FDA approved and commercially available. Their use in this study is investigational. Up to 36 patients will take part in this multicenter study. Up to 36 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosis of low-grade indolent lymphomas Stage I-II. Patients with multiple skin lesions will be eligible provided that the skin is the only site of involvement.
2. Histology includes Indolent cluster of differentiation antigen 20 (CD20)+ lymphomas including: Follicular lymphoma, Extranodal marginal lymphoma of MALT type, Nodal Marginal zone B-cell lymphoma (+/- monocytoid cells), and Splenic marginal B-cell lymphoma (+/- villous lymphocytes).
3. Signed Informed Consent.
4. Age >/= 18 years.
5. Pre-study Zubrod performance status of 0, 1, or 2.
6. Acceptable hematologic status within two weeks prior to patient registration, including: absolute neutrophil count ([segmented neutrophils + bands] x total WBC) >/= 1, 500/mm^3, total lymphocyte count </= 5,000/mm^3 and platelet counts >/= 100,000/mm^3.
7. Female patients who are not pregnant or lactating.
8. Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician, however abstinence is not an acceptable method).
9. Patients determined to have < 25% bone marrow involvement with lymphoma within six weeks of registration (define measurement of a bone marrow aspirate or biopsy).
10. Patient should have at least one lesion measuring >/= 1.5 cm in a single dimension. Measurable cutaneous lesions are allowed.

Exclusion Criteria:

1. Presence of central nervous system (CNS) lymphoma.
2. Patients with HIV or AIDS-related lymphoma.
3. Patients with pleural effusion.
4. Patients with abnormal liver function: total bilirubin > 2.0 mg/dL.
5. Patients with abnormal renal function: serum creatinine > 2.0 mg/dL.
6. Patients who have received prior external beam radiation therapy to > 25% of active bone marrow (involved field or regional).
7. Impaired bone marrow reserve as indicated by < 15% bone marrow cellularity
8. Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives.
9. Major surgery, other than diagnostic surgery, within four weeks.
10. Evidence of transformation in the latest biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-06; Primary Completion 2015-04 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Samaniego, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 12, 2006 to May 08, 2009. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Zevalin: Ibritumomab Tiuxetan (Zevalin): 111In Zevalin (5 mCi of ^111In, 1.6 mg of Ibritumomab Tiuxetan) intravenous (IV) over 10 minutes on Day 1; 90Y Zevalin 0.3 or 0.4 mCi/kg IV over 10 minutes on Day 8. Rituximab: 250 mg/m^2 IV over 4-6 Hours on Days 1 and 8 prior to the administration of 111In Zevalin and 90Y Zevalin, respectively.
Period: Overall Study
Arm/Group | Zevalin
Started | 31
Completed | 30
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zevalin
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 60 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR defined as the percentage of number of complete response (CR), complete response unconfirmed (CRu) or partial response (PR) in patients treated using International Working Group (IWG) revised response criteria for Malignant Lymphoma. ORR to therapy is evaluated after three months using radiographic and clinical parameters to assess response. CR: Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms. CRu: A residual lymph node mass greater than 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the products of the greatest diameters (SPD). Individual nodes that were previously confluent must have regressed by more than 75% in their SPD compared to the original mass and indeterminate bone marrow. PR: ≥ 50% decrease in SPD of the six largest dominant nodes or nodal masses. No increase in the size of other nodes, liver or spleen and no new sites of disease.
Time Frame: Up to 5 years; Evaluation at 3-month intervals during Year 1, then every 6 months to Year 4. The median follow-up was 56 months for censored observations.
Measure: Number; unit: Percentage of Participants
Arm/Group | Zevalin
Number analyzed (Participants) | 31
Percentage of Participants
  Complete Response | 67.7
  Complete Response Unconfirmed | 29.0
  Partial Response | 3.3

2. Secondary Outcome: Progression Free Survival (PFS) Rate at 3 Years
Description: PFS measured, in a responder, from the date when a CR, CRu or PR is first noted to the first date at which progressive disease is observed or death. An ongoing PFS interval occurs when there is a responder for whom progressive disease has not been noted. Progression of disease defined as enlargement of liver/spleen, new sites observed, new or increased lymph nodes or lymph node masses, or reappearance of bone marrow.
Time Frame: Evaluation at 3-month intervals during the first year and then every 6 months until year 3
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Zevalin
Number analyzed (Participants) | 31
Proportion of participants
  Male | 0.62 [0.40 to 0.95]
  Female | 0.89 [0.75 to 1.00]

ADVERSE EVENTS:
Time Frame: Adverse events collected during treatment period including time from first Rituxan infusion (through Day 8) up to 12 weeks following Zevalin infusion.
Arm/Group | Zevalin
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin (N=31)
PERFORATION, GI (Gastrointestinal disorders) | 1 (1) — Small bowel perforation
DEATH (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin (N=31)
ABDOMEN PAIN (Gastrointestinal disorders) | 2 (2)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 2 (2)
ALLERGIC RHINITIS (Immune system disorders) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 1 (1)
BLADDER INFECTION (Infections and infestations) | 1 (1)
BLURRED VISION (Eye disorders) | 4 (4)
BRUISING (Injury, poisoning and procedural complications) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 4 (4)
COUGH (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 4 (4)
DIZZINESS (Nervous system disorders) | 4 (4)
DRY EYE (Eye disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EDEMA: HEAD AND NECK (General disorders) | 1 (1)
EDEMA: LIMB (General disorders) | 4 (4)
FATIGUE (General disorders) | 19 (19)
FEVER WITHOUT NEUTROPHIL INCREASE (Investigations) | 4 (4)
HEADACHE (Nervous system disorders) | 3 (3)
HEARTBURN (Gastrointestinal disorders) | 1 (1)
HEMOGLOBIN INCREASE (Investigations) | 12 (12)
HEMORRHAGE, PULMONARY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTION UNKNOWN (Infections and infestations) | 2 (2)
INFECTION WITHOUT NEUTROPHIL INCREASE (Infections and infestations) | 2 (2)
INSOMNIA (Psychiatric disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 19 (19)
MUSCLE SPASM (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 8 (8)
NEUROPATHY: SENSOR (Nervous system disorders) | 8 (8)
NEUTROPHILS CHANGE (Absolute neutrophil count (ANC)) (Investigations) | 21 (21)
PAIN (General disorders) | 1 (1)
PAIN (ABDOMEN NOS) (Gastrointestinal disorders) | 1 (1)
PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN (HEAD/HEADACHES) (Nervous system disorders) | 2 (2)
PAIN (JOINT) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN (MUSCLE) (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN PELVIC (Reproductive system and breast disorders) | 1 (1)
PERFORATION, GI (Gastrointestinal disorders) | 1 (1)
PLATELETS, DECREASE (Investigations) | 21 (21)
PROPTOSIS/Enophthalmos (Eye disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (1)
REDNESS OF EYES (Eye disorders) | 2 (2)
RIGORS/CHILLS (General disorders) | 1 (1)
SWEATING (General disorders) | 3 (3)
THROMBOSIS/THROMBUS (Vascular disorders) | 1 (1)
TINNITUS (Eye disorders) | 1 (1)
VAGINAL BLEEDING (Reproductive system and breast disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No